CLINICAL TRIAL: NCT05971056
Title: A Natural Experiment of Providing Cancer Care Closer to Home for Patients With Multiple Myeloma
Brief Title: Providing Cancer Care Closer to Home for Patients With Multiple Myeloma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202306162
Record Dates: First submitted 2023-07-20; First posted 2023-08-02 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma
Keywords: access to care; travel burden; financial toxicity; patient satisfaction
MeSH Terms: conditions — Multiple Myeloma; Financial Stress; Patient Satisfaction | interventions — Patient Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care transition (Experimental): -At baseline, the participant and the provider will make a decision on if the participant will transfer care to a satellite location.
  Interventions: Other: Care transition
- No care transition (Active Comparator): -At baseline, the participant and the provider will make a decision on if the participant will transfer care to a satellite location.
  Interventions: Other: No care transition

INTERVENTIONS:
Other: Care transition — Cancer care is transitioned to a satellite site.
  Arms: Care transition
Other: No care transition — Cancer care is not transitioned to a satellite site.
  Arms: No care transition

SUMMARY:
There is very limited data on the utilization of National Cancer Institute Comprehensive Cancer Center (NCI-CCC) satellite sites in general. Of what is available, most is in regards to providing chemotherapy at facilities closer to patients' home. These "satellite chemotherapy infusion centers", typically community-based treatment locations at community hospitals/facilities, freestanding clinics, or mobile units, are reported to be well liked by patients who utilize their services and reduce their travel times and expenses. In these studies patients still remained in the care of their current provider and site and are required to travel to the site for clinical visits and other appointments. It is currently unknown if patients are willing to transfer their care to a different provider to alleviate travel burden. In addition, although increased travel burden has been lower quality of life in cross-sectional studies, no data exists suggesting that these reducing travel burden can improve these outcomes intra-patient, to the knowledge of the investigators.

The patient roles of the multiple myeloma clinical providers at the Siteman primary location have grown in recent years. The providers have determined a need to refer some patients to the satellite sites to relieve congestion at the site while also hopefully improving the clinical experience for those patients. This study is a natural experiment of this process.

ELIGIBILITY:
Eligibility Criteria

* At least 18 years old
* Diagnosed with multiple myeloma
* Receiving care from a provider within the Division of Oncology at the primary Siteman Cancer Center site
* Resides within the catchment area of a Siteman Cancer Center satellite site
* Able to read, speak, and understand English
* Willing to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible participants who successfully transfer to the provider at a satellite location | At time of transfer decision (day 1)

SECONDARY OUTCOMES:
Types of candidacy that providers use for transfer of care to satellite sites | At time of transfer decision (day 1)
  Qualitative data collection
Treatment burden of participants as measured by the Modified Treatment Burden Questionnaire | Through completion of follow-up (estimated to be 6 months)
  * Explore differences in participant experience between those that elect to transfer to a satellite site and those who decline to transfer.
  * The Modified Treatment Burden Questionnaire will be completed at baseline (time of transfer decision) and again approximately 6 months later. There are 3 questions with answers ranging from 0 (not a problem) to 10 (big problem). The higher the score the more treatment burden the participant experienced.
Satisfaction of with participant-provider interactions as measured by the Questionnaire on the Quality of Physician-Patient Interaction | Through completion of follow-up (estimated to be 6 months)
  * Explore differences in participant satisfaction between those that elect to transfer to a satellite site and those who decline to transfer.
  * The Questionnaire on the Quality of Physician-Patient Interaction will be completed at baseline (time of transfer decision) and again approximately 6 months later. There are 14 questions with answers ranging from 1 (do not agree) to 5 (I fully agree). The higher the score the higher the quality of the physician-patient interactions.
Financial toxicity of participants as measured by the Comprehensive Score for Financial Toxicity | Through completion of follow-up (estimated to be 6 months)
  * Explore differences in participant financial toxicity between those that elect to transfer to a satellite site and those who decline to transfer.
  * The Comprehensive Score for Financial Toxicity will be completed at baseline (time of transfer decision) and again approximately 6 months later. There are 11 questions with answers ranging from 0 (not at all) to 4 (very much). The higher the score the less financial toxicity the participant experienced.
Participant rationales for opting to transfer to a satellite site or maintain care at their usual site. | Through completion of follow-up (estimated to be 6 months)
  A sample of 20 patients, approximately 10 who decided to transfer and 10 who declined, will be surveyed in regards to the reason(s) for their decision as part of a sub-study. Patients who were not enrolled in the prospective portion of the study, either due to declining or not approached, will be allowed to enroll in the sub-study as long as they were offered the ability to transfer to a satellite site by their provider.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fiala, Ph.D., MSW, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu